CLINICAL TRIAL: NCT07337304
Title: Comparative Effects of Single vs. Multiple-Set Resistance Training on Neuromuscular Performance and Muscle Morphology in Sedentary Men
Brief Title: Single vs. Multiple-Set Resistance Training in Sedentary Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ilgin Ali Coskun, Researcher, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INU-RT-SSMS-01
Record Dates: First submitted 2025-12-14; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Resistance Training Adaptation; Sedentary Lifestyle; Neuromuscular Adaptations
Keywords: Resistance training; Single-set training; Multiple-set training; Neuromuscular performance; Muscle morphology; Sedentary men
MeSH Terms: conditions — Sedentary Behavior | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three parallel groups: single-set resistance training, multiple-set resistance training, or a non-exercising control group. All groups were followed concurrently throughout the intervention period.
Masking Description: This study was conducted as an open-label trial. Due to the nature of the exercise interventions, neither participants nor investigators were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-Set Resistance Training (Experimental): Participants performed a supervised resistance training program consisting of one set per exercise. Training was conducted at moderate intensity using standard resistance exercises targeting major muscle groups.
  Interventions: Behavioral: Resistance Training
- Multiple-Set Resistance Training (Experimental): Participants performed a supervised resistance training program consisting of multiple sets per exercise. Exercise selection, intensity, and training frequency were comparable to the single-set group.
  Interventions: Behavioral: Resistance Training
- Control Group (No Intervention): Participants did not participate in any structured exercise training program and were instructed to maintain their usual daily activities throughout the study period.

INTERVENTIONS:
Behavioral: Resistance Training — A structured and supervised resistance training program performed at moderate intensity using free weights and resistance machines.
  Arms: Multiple-Set Resistance Training; Single-Set Resistance Training

SUMMARY:
This study aimed to compare the effects of single-set versus multiple-set resistance training on neuromuscular performance and muscle morphology in sedentary men. Participants were randomly assigned to a single-set training group, a multiple-set training group, or a non-training control group. The intervention consisted of a structured resistance training program performed over a defined training period, while the control group maintained their usual lifestyle without structured exercise. Neuromuscular performance outcomes included maximal strength and functional performance measures, and muscle morphology was assessed using appropriate imaging and anthropometric methods. The findings of this study are intended to contribute to the understanding of optimal resistance training volume for improving neuromuscular adaptations in previously untrained individuals.

DETAILED DESCRIPTION:
This randomized controlled trial was designed to investigate the effects of resistance training volume on neuromuscular performance and muscle morphology in sedentary adult men. Participants with no regular resistance training history were recruited and randomly allocated into three groups: a single-set resistance training group, a multiple-set resistance training group, and a non-training control group.

Both training groups participated in a supervised resistance training program targeting major muscle groups. The single-set group performed one set per exercise, while the multiple-set group performed multiple sets per exercise, using comparable exercise selection, intensity progression, and rest intervals. Training sessions were conducted at a consistent weekly frequency over the intervention period. The control group did not engage in any structured exercise program and was instructed to maintain their habitual daily activities throughout the study.

Neuromuscular performance was evaluated using maximal strength and functional performance assessments conducted before and after the intervention period. Muscle morphology outcomes were assessed using standardized measurement techniques appropriate for evaluating changes in muscle size and structure. All assessments were performed by trained personnel following standardized protocols.

The primary objective of the study was to compare the magnitude of neuromuscular and morphological adaptations between single-set and multiple-set resistance training protocols in previously untrained individuals. Secondary objectives included comparing both training interventions with a non-training control condition. The results of this study aim to provide evidence-based insight into the effectiveness of different resistance training volumes for improving neuromuscular adaptations in sedentary populations.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged between 18 and 40 years
* Sedentary lifestyle (no structured resistance training in the previous 6 months)
* Apparently healthy, with no known cardiovascular, metabolic, or musculoskeletal disorders
* Ability to participate in resistance training exercise
* Willingness to provide written informed consent

Exclusion Criteria:

* Participation in regular resistance or structured exercise training within the past 6 months
* History of musculoskeletal injury or surgery that could limit exercise performance
* Presence of cardiovascular, neurological, or metabolic disease
* Use of medications or supplements known to affect muscle function or performance
* Any condition deemed unsafe for participation by the investigators

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Maximal Muscle Strength (1RM) | Baseline and Week 8
  Change in maximal muscle strength assessed by one-repetition maximum (1RM) testing for major upper- and lower-body exercises.

SECONDARY OUTCOMES:
Muscle morphology | Baseline and Week 8
  Changes in muscle morphology assessed using fat-free mass, body fat percentage, and limb circumference measurements.
Vertical Jump Height | Baseline and Week 8
  Change in vertical jump height assessed using a standardized countermovement jump test to evaluate lower-body explosive power.
20-m Sprint Time | Baseline and Week 8
  Change in 20-meter sprint time assessed using electronic timing gates to evaluate short-distance sprint performance.
Handgrip Strength | Baseline and Week 8
  Change in maximal handgrip strength assessed using a calibrated handgrip dynamometer to evaluate upper-body isometric strength.
Estimated VO₂max | Baseline and Week 8
  Change in estimated maximal oxygen uptake derived from performance in the Yo-Yo Intermittent Recovery Test Level 1.
Perceived Exertion (OMNI-RES) | Baseline and Week 8
  Change in perceived exertion assessed using the OMNI-Resistance Exercise Scale during resistance training sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Faculty of Sport Sciences, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No